CLINICAL TRIAL: NCT00975169
Title: Association Study of Genetic Polymorphisms of Candidate Genes With Thiazolidinedione-Related Peripheral Edema and Drug Responsiveness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Tien-Jyun Chang, National Taiwan Univerisity Hospital
Other Study IDs: 200902005R
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TZDs User

SUMMARY:
According to the above evidence, though the exact mechanism contributing to the Thiazolidinediones (TZDs) associated peripheral edema is still unclear, the investigators hypothesize that the genetic variations of certain candidate genes involved in peroxisome proliferator-activated receptor (PPAR) gamma itself and PPAR gamma-regulated genes may contribute to TZDs-associated peripheral edema. Therefore, the investigators plan to conduct a case-control study to test the association between single nucleotide polymorphisms (SNPs) in certain candidate genes and TZDs related peripheral edema.

A large fraction of individuals, both with type 2 diabetes (38-41) or who are at risk for type 2 diabetes, do not respond to TZD therapy. In individuals with type 2 diabetes, non-response has not been carefully characterized, but data from studies in at-risk individuals suggests that a lack of improvement in insulin sensitivity (Si) may account for the lack of response to TZD therapy. In the Troglitazone In the Prevention Of Diabetes (TRIPOD) study, around 30% of treated women did not show an improvement in Si; they gained no protection from type 2 diabetes when compared with the placebo group. Assessment of baseline clinical and physiologic measurements revealed similar levels of adiposity, fasting glucose and insulin, Si and β-cell function, fasting lipids, contraceptive use, and compliance with study medication between responders and nonresponders, suggesting that these measures do not predict TZD response.

The adipose tissue-derived hormone adiponectin improves insulin sensitivity and its circulating levels are decreased in obesity induced insulin resistance. In ob/ob mice lacking adiponectin, the ability of PPARγ agonists, TZDs, to improve glucose tolerance is diminished. It implied that adiponectin is an important contributor to PPARγ-mediated improvements in glucose tolerance through mechanisms that involve the activation of the AMPK pathway. On the other hand, it has been shown that FOXO1 repressed PPARγ1 and γ2 promoters in primary adipocytes. It has also been reported that peroxisome proliferators activated receptor-γ coactivator-1α (PGC-1α) gene expression in brown and white adipocytes is a direct target of TZDs and activators of retinoid X receptor (RXR). Taken together, both FOXO1 and PGC-1α potentially played important roles on the antidiabetic action of TZDs.

In summary, though TZDs have been widely used in patients with type 2 diabetes mellitus, some of patients experienced TZD-related peripheral edema and some of patients had no good responsiveness to TZDs. The underlying contributing factors and molecular mechanisms have not been clearly elucidated. In this study, the investigators will identify the contributing factors of TZD-related peripheral edema and responsiveness to TZDs. The investigators will also identify the association of single nucleotide polymorphisms (SNPs) of certain candidate genes with TZD related peripheral edema and responsiveness to TZDs. It may identify some clinical and pharmacogenetic factors to predict the occurrence of TZD-related edema and the responsiveness to TZDs.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of DM and with use TZDs

Exclusion Criteria:

* Patients with the diagnosis of congestive heart failure
* Liver cirrhosis (according to abdominal echo)
* Renal insufficiency (Cr ≥ 1.7 mg/dL)
* Patient with concomitant use of insulin, and/or diuretics before TZDs were excluded
* Pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: TZDs User, no insulin; CHF, according to New York heart Association III-V, liver cirrhosis or renal insufficiency (Cr ≥ 1.7 mg/dL) before initiation of treatment with TZDs will be excluded.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
we plan to conduct a case-control study to test the association between single nucleotide polymorphisms (SNPs) in certain candidate genes and TZDs related peripheral edema | 34 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tien-Jyun Chang, Ph D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Internal Medicine, National Taiwan University Hospital, Taipei, Taiwan